CLINICAL TRIAL: NCT06349941
Title: Implementing a Home-based Cardiac Rehabilitation Program Among Rural Patients With Heart Failure
Brief Title: Home-based Cardiac Rehabilitation in Heart Failure
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ambarish Pandey, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2023-0745
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure
Keywords: telehealth; heart failure; rural; cardiac rehabilitaion
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Movn cardiac rehabilitation (Experimental): Cardiac rehabilitation delivered through Movn app through the use of mHealth.
  Interventions: Device: Movn app
- Attention Control (Active Comparator): This group will receive a wearable device for step count tracking and will get periodic check ins to minimize differential attention between groups. They will not receive an exercise plan.
  Interventions: Device: Accelerometer

INTERVENTIONS:
Device: Movn app — Participants will have 12-week home-based exercise program delivered via a commercially available home-based cardiac rehabilitation platform called Movn. The plan includes an accelerometer, blood pressure scale, and mobile application.
  Other Names: Cardiac Rehabilitation
  Arms: Movn cardiac rehabilitation
Device: Accelerometer — Participants will receive a FitBit for monitoring of physical function.
  Other Names: FitBit
  Arms: Attention Control

SUMMARY:
This study evaluates a mobile health (mHealth) home-based cardiac rehabilitation program for patients with heart failure. We will stratify randomization between rural and urban populations, with the goal to assess implementation of cardiac rehabilitation across these two geographic areas. . The study will randomize 332 patients with heart failure (ejection fraction ≥35%) who are not eligible for center-based rehabilitation to either a 12-week mHealth cardiac rehabilitation program or an attention control group, with outcomes measured over 6 months using a composite endpoint of mortality, hospitalizations, and quality of life. We will then assess the implementation of the intervention.

DETAILED DESCRIPTION:
Background and Significance:

Rural communities in the United States experience a disproportionate burden of cardiovascular disease and associated adverse outcomes, with recent epidemiological data demonstrating a widening mortality gap compared to urban populations. These disparities are particularly pronounced in cardiovascular care delivery, where rural-residing adults demonstrate significantly lower rates of guideline-directed therapies for coronary heart disease, heart failure, and stroke. Among the most substantial gaps identified is the utilization of cardiac rehabilitation services, with total participation among Medicare beneficiaries reaching only 5% in rural areas. This disparity is compounded by the intersection of multiple risk factors including reduced access to healthcare services, lower socioeconomic status, and geographic barriers to specialized care.

The emergence of telemedicine platforms presents a novel opportunity to address these healthcare access disparities through innovative service delivery models. The COVID-19 pandemic has catalyzed the adoption of digital health technologies, with telemedicine visits among rural Medicare beneficiaries increasing nearly 100-fold between 2019 and 2020. Concurrent improvements in rural broadband access, with over 70% of rural adults reporting home broadband availability in 2021, have created an infrastructure foundation supporting telehealth interventions. Mobile health (mHealth) interventions have demonstrated efficacy in cardiovascular care through patient monitoring, medication adherence support, and risk factor management, with preliminary evidence suggesting effectiveness in reducing rehospitalizations and increasing patient participation in cardiac rehabilitation programs.

Study Design and Methodology:

This investigation employs a randomized, open-label, Type 1 hybrid effectiveness-implementation trial design to evaluate the efficacy and implementation characteristics of an mHealth-enabled home-based cardiac rehabilitation program. The study will enroll 332 adult participants with recent hospitalization for heart failure with ejection fraction ≥35%, stratified with 70% recruitment from rural hospitals and 30% from urban centers to enable comparative analysis of implementation challenges across geographic settings. Participants will be randomized in a 1:1 ratio to receive either the mHealth cardiac rehabilitation intervention or attention control, with outcomes assessed over a 6-month follow-up period.

Intervention Components:

Participants randomized to the mHealth cardiac rehabilitation group receive a comprehensive remote monitoring kit delivered via overnight shipping, containing a wireless blood pressure monitor, resistance bands, and a wearable monitor. These hardware components integrate with the Movn Health platform, which participants access through a smartphone application offering both synchronous and asynchronous features including real-time video consultations with exercise coaches, exercise videos for self-directed sessions, one-to-one messaging capabilities, and automatic data synchronization from all monitoring devices.

The 12-week cardiac rehabilitation program implements a multi-domain physical rehabilitation approach. The intervention begins with a comprehensive assessment evaluating exercise capacity and safety requirements. Each participant follows a personalized exercise regimen.

Participants in the attention control group receive a FitBit device for activity monitoring and step count tracking, along with bi-weekly telephone calls throughout the 12-week intervention period to minimize contact differential between study arms. These telephone interactions focus on general health discussions without providing specific exercise counseling or rehabilitation guidance.

Outcome Measures and Assessment:

The primary endpoint employs a composite hierarchical outcome structure analyzed using a win-ratio methodology, incorporating all-cause mortality, time to first heart failure hospitalization, total heart failure hospitalizations, and a 5-point difference in quality of life assessed by the Kansas City Cardiomyopathy Questionnaire. This analytical approach provides a comprehensive evaluation of intervention effectiveness across multiple clinically relevant domains while accounting for the relative importance of mortality and morbidity outcomes.

Secondary endpoints include individual components of the primary composite outcome, physical activity levels measured through FitBit-recorded daily step counts, and general health-related quality of life assessed using the EuroQol 5 Dimension 5 Level instrument. Additional secondary measures encompass mental health parameters evaluated through the Patient Health Questionnaire-9, Generalized Anxiety Disorder-7 scale, and the Physical Activity Scale for the Elderly.

The study incorporates comprehensive implementation outcome assessment using the RE-AIM framework, evaluating Reach through the number of eligible participants receiving the intervention, Effectiveness through perceived relative advantage and observed outcomes, Adoption through adherence rates and contextual factors, Implementation through fidelity measures and cost analysis, and Maintenance through persistence and discontinuation rates. A sequential mixed-methods approach will conduct semi-structured interviews with 12 clinicians across all sites and 36 patients across study arms to evaluate acceptability, preferences, and contextual factors influencing implementation effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* History of hospitalization for acute heart failure with ejection fraction ≥ 35%
* Ability to participate in telemedicine visits
* Access to smartphone or device capable of running the mHealth application
* Willingness to participate in home-based cardiac rehabilitation program

Exclusion Criteria:

* Heart failure with reduced ejection fraction (ejection fraction < 35%)
* Inability to participate in physical exercise or cardiac rehabilitation due to medical contraindications
* Inability to provide informed consent
* Lack of access to required technology (smartphone, internet connectivity)
* Life expectancy less than 6 months
* Inability to participate in telemedicine visits or remote monitoring
* Current participation in another cardiac rehabilitation program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Composite Hierarchical Endpoint | 6 months.
  A composite outcome incorporating all-cause mortality, time to first heart failure hospitalization, total heart failure hospitalizations, and a 5-point difference in disease-specific quality of life score as assessed by the Kansas City Cardiomyopathy Questionnaire (KCCQ). The KCCQ ranges from 0-100, where 0 indicates worst quality of life and 100 indicates best quality of life.

SECONDARY OUTCOMES:
Physical Activity Level | Continuously measured over 6 months.
  Daily Step Count
General Health-Related Quality of Life | Baseline, 3 months, and 6 months
  Change in general health-related quality of life assessed using the EuroQol 5 Dimension 5 Level (EQ-5D-5L) instrument. The EQ-5D-5L uses a descriptive system to measure health-related quality of life across five key dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on five levels of severity-ranging from no problems (Level 1) to extreme problems or inability to function (Level 5). A respondent's answers generate a five-digit health state profile that reflects their unique combination of responses (e.g., 12345), representing one of 3,125 possible health states. This descriptive system enables consistent and standardized assessment of an individual's health status.
Implementation Outcomes | Assessed at 3 and 6 months.
  Assessment of the implementation of the cardiac rehabilitation program using mixed methods evaluation.
Depressive Symptoms | Baseline, 3 months, and 6 months
  Change in mental health parameters assessed using the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 ranges from 0 to 27, with higher scores indicating more severe depressive symptoms.
Anxiety Symptoms | Baseline, 3 months, and 6 months
  Change in anxiety symptoms assessed using the Generalized Anxiety Disorder-7 (GAD-7) scale. Total scores range from 0 to 21, with higher scoes indicating more severe anxiety symptoms.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor Scott and White Health System, Dallas, Texas